CLINICAL TRIAL: NCT04144530
Title: MRI Repository for Acute Stroke Clinical and Research Applications
Status: Withdrawn | Type: Observational
Why Stopped: study did not start by logistic reasons
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00228775
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is one of the leading causes of death and long-term disability. A major unresolved problem in MRI-based stroke assessment is to relate image features to brain function in a way that can properly guide stratification for treatment and rehabilitation. This requires extracting meaningful and reproducible models of brain function from stroke images, a daunting task severely hindered by the great variability of lesion frequency and pattern. Large datasets are imperative to uncover possible lesion-function relationships.

In this project the investigators will create a large database of acute strokes MRIs. The investigators will retrospectively archive an estimated 3,000 MRIs of patients with acute stroke, acquired at the Johns Hopkins Hospital, 2009-2019. This dataset will include 1.5 and 3 Tesla scans, diverse protocols and sequences (e.g., diffusion and perfusion weighted images (DWI/b0, PWI), T1, T2, FLAIR, susceptibility weighted images), with typical clinical low voxel resolution (4-7 mm3). Lesions will be initially delineated on DWI/b0, the most informative MRI sequence for acute stroke. After anonymization and defacing, two trained evaluators will perform the manual lesion segmentation. Two expert neuroradiologists will create consensual structured radiological reports with information about stroke type and location according to different criteria (e.g., 34 brain structures and 11 vascular territories). The investigators will also archive structured information from discharge (demographics, laboratory, and neurological evaluation of patients, including NIH stroke scale and modified Rankin scale, mRS), as well as the 90-days follow-up mRS.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted at Hopkins Stroke center with the diagnosis of acute brain stroke

Exclusion Criteria:

* Not performed MRI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted at Hopkins Stroke center with the diagnosis of acute brain stroke
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Demographic and clinical data obtained via chart review | 1 year
  This is a hospital based retrospective collection of data for acute stroke from a ten-year period retrospective review of participant charts.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia V Faria, MD, PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the database public in sharing neuroimaging platforms after anonymization, including defacing.
Supporting Information: Analytic Code